CLINICAL TRIAL: NCT06735053
Title: Experimental Study on the Impact of a Virtual Reality-Based Physiotherapy Program as a Complement to a Conventional Physiotherapy Program in Patients With Moderate to Severe Multiple Sclerosis
Brief Title: Impact of Virtual Reality Physiotherapy on Multiple Sclerosis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Marina Castel Sánchez, PhD, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24/765-EC_P
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; virtual reality
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): The intervention group will carry out a physiotherapy program using virtual reality and conventional treatment for 10 weeks. They will receive 2 weekly treatment sessions of 60 minutes distributed in 45 minutes of physiotherapy using the virtual reality based device (Dynamics VR) following a therapeutic protocol where patients will have exercise sessions based on the theory of motor learning with upper limb and trunk work including fine motor and gross motor exercises, trunk control and postural control exercises, increasing the level of demand or difficulty of the exercises as the weeks go by. Additionally, they will receive a complement of 15 minutes of treatment with conventional physiotherapy directed to the specific needs of each patient.
  Interventions: Other: Virtual Reality group
- Placebo Virtual reality group (Placebo Comparator): The control group will carry out a conventional physiotherapy program for 10 weeks in which they will receive 2 weekly treatment sessions of 60 minutes distributed in 45 minutes of physiotherapy and 15 minutes of treatment with online virtual reality placebo.
  Interventions: Other: Placebo virtual reality group

INTERVENTIONS:
Other: Virtual Reality group — Virtual reality group will perform online reality-based device following a therapeutic protocol supervised by a physiotherapist in which the level of demand will be adjusted to the patient's evolution. This programme provides a gamified and challenging online environment to enhance motor learning and induce sensorimotor adaptations. Additionally, they will receive conventional physiotherapy approach, oriented to the specific objectives of each patient, aiming to normalize tone, activate weakened muscles, facilitate movement, recover sensitivity, and compensate for functional deficits. Additionally, global kinesitherapy, motor coordination exercises, pedalier, vibration therapy (vibrosphere®), and analgesic electrotherapy will be performed if necessary.
  Arms: Virtual Reality group
Other: Placebo virtual reality group — The control group will undergo a conventional physiotherapy program based on the normalization of tone, activation of weakened muscles and facilitation of normal movement, recovery of alterations in sensitivity, and compensation of lost functional deficits. In addition, global kinesitherapy exercises will be performed on a stretcher, motor coordination exercises, pedalier, vibration therapy (vibrosphere ®) and analgesic electrotherapy if necessary. Finally, in order to minimize the differences between the control and intervention groups, the participants of the control group will watch a 15-minute generic 2D video freely accessible on the Youtube platform from the VR glasses, without specific software.
  Arms: Placebo Virtual reality group

SUMMARY:
The goal of this clinical trial is to learn if virtual reality combined with conventional physiotherapy intervention works to treat moderate to severe multiple sclerosis persons. The main questions it aims to answer are:

* Does the application of a virtual reality-based program along with conventional physiotherapy produces improvements compared to the application of conventional physiotherapy and placebo virtual reality in motor aspects of patients with multiple sclerosis?
* Does the application of a virtual reality-based program along with conventional physiotherapy produces improvements compared to the application of conventional physiotherapy and placebo virtual reality in cognitive aspects of patients with multiple sclerosis

Researchers will compare a virtual reality-based program along with conventional physiotherapy with a placebo virtual reality to see if virtual reality improve motor and cognitive aspects of multiple sclerosis.

Participants will:

* Visit the clinic twice a week for 10 weeks to receive a 1-hour session of virtual reality and conventional physiotherapy.
* Be assessed using various scales and questionnaires at three different times: at the start of the study, at the end of the treatment, and 4 weeks after the study ends.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis based on McDonald criteria, with an evolution time of more than two years.
* All patients with Multiple Sclerosis are included according to the Kurtzke Multiple Sclerosis Disability Status Scale (EDSS) (ANNEX II) with a score greater than or equal to 6.5 (Need of two types of support to walk -two canes, walker...- about 20 meters without resting).
* Stable medical treatment for at least six months prior to intervention.
* Absence of cognitive impairment, with ability to understand instructions and to obtain a score equal to or greater than 24 on the Minimental Test.

Exclusion Criteria:

* Diagnosis of another neurological disease or musculoskeletal disorder other than MS.
* Diagnosis of any cardiovascular, respiratory or metabolic disease, or other conditions that may interfere with this study.
* To have suffered an exacerbation or hospitalization in the last 3 months before starting the assessment protocol, nor during the therapeutic intervention process.
* To have received a course of steroids, intravenously or orally, 6 months prior to the start of the assessment protocol and within the intervention period of the study duration.
* Visual disturbances not corrected by ocular devices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue impact as measured with Modified Fatigue Impact Scale (MFIS) | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  Modified Fatigue Impact Scale is a self-report questionnaire designed to assess the impact of fatigue on patients with multiple sclerosis (MS). It evaluates how fatigue affects physical, cognitive, and psychosocial functioning on daily life in MS patients. The MFIS consists of 21 items divided into three subscales: physical, cognitive, and psychosocial. Higher scores indicate a greater impact of fatigue. The total score is the sum of all item scores, with subscale scores calculated separately.
  The administration time is approximately 5-10 minutes. It is typically self-administered, but can be conducted as an interview if necessary.

SECONDARY OUTCOMES:
Change in Physical and psicological impact of Multiple Sclerosis on patients'life measured with Multiple Sclerosis Impact Scale (MSIS-29) | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  MSIS-29 is patient-reported outcome measure designed to assess the physical and psychological impact of multiple sclerosis on patients' lives. It consists of 29 items divided into two subscales:
  * Physical Impact (20 items): Evaluates the physical limitations and challenges faced by MS patients.
  * Psychological Impact (9 items): Assesses the emotional and cognitive effects of MS.
  Each item is rated on a scale, with higher scores indicating a greater impact of MS. The total score is the sum of the physical and psychological subscale scores. The administration Time is approximately 10-15 minutes. It can be self-administered or conducted as an interview.
Change in manual dexterity and fine motor skills | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be measured using the Purdue Pegboard TEST (PPT). It is a performance-based assessment used to measure manual dexterity and fine motor skills. Assesses fine motor skills and coordination of the fingers, hands, and arms. The test involves a rectangular board with two sets of 25 holes and four concave cups at the top. Participants are asked to place small metal pegs into the holes as quickly as possible. The test includes five subtests: right hand, left hand, both hands, right + left + both hands (a calculated score), and an assembly task. Each subtest is timed, typically 30 seconds for the hand tasks and 60 seconds for the assembly task. The administration time is approximately 5-10 minutes. It will be conducted by a test administrator. The participant is seated during the test.
Change in gross motor manual dexterity | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be evaluated through the Box and Block Test (BBT). It is designed to assess gross manual dexterity by measuring the ability to move small blocks from one compartment to another.The test involves a rectangular box divided into two equal compartments by a partition. One hundred and fifty small wooden blocks (2.5 cm each) are placed in one compartment. Participants are instructed to move as many blocks as possible, one at a time, from one compartment to the other within a 60-second period. The score is the number of blocks successfully transferred within the time limit. Higher scores indicate better manual dexterity. The administration time is approximately 2-5 minutes. The test will be administered with the participant seated at a table, and it will be conducted by a clinician or researcher.
Change in functional independence to perform activities of daily living | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be assessed using The Barthel Index (BI). It assesses the ability to perform activities of daily living (ADLs) independently. Evaluates the degree of assistance required by an individual to perform 10 basic ADLs, including feeding, bathing, grooming, dressing, bowel and bladder control, toilet use, transfers (e.g., from chair to bed), mobility, and stair climbing.
  The index consists of 10 items, each scored on a scale that reflects the level of independence. The total score ranges from 0 to 100, with higher scores indicating greater independence.
  Each activity is scored based on the amount of assistance required, with possible scores of 0 (dependent), 5 (needs some help), or 10 (independent) for most items. The total score is the sum of the individual item scores.The administration time is approximately 5-10 minutes.
  It can be administered through direct observation, patient self-report, or interviews with caregivers.
Change in the ability to perform instrumental activities of daily living | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be measured with the Lawton-Brody Instrumental Activities of Daily Living (IADL) Scale. It is a tool used to assess an individual's ability to perform complex daily activities necessary for independent living. Measures the ability to perform instrumental activities of daily living, which are more complex than basic self-care tasks.
  The scale includes 8 items that assess activities such as using the telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and handling finances.
  Each item is scored based on the level of independence, with a total score ranging from 0 (low function, dependent) to 8 (high function, independent). For men, the score ranges from 0 to 5 to avoid gender bias.
  The administration time is approximately 10-15 minutes. It can be administered through an interview or a written questionnaire, with responses provided by the patient or a caregiver familiar with the patient's abilities.
Change in cognitive function | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be assessed with the Montreal Cognitive Assessment (MoCA). It evaluates multiple cognitive domains to provide a comprehensive overview of an individual's cognitive abilities.
  The MoCA includes tasks that measure attention and concentration, executive functions, memory, language, visuospatial skills, conceptual thinking, calculations, and orientation.
  The test is scored out of 30 points, with higher scores indicating better cognitive function. A score of 26 or above is generally considered normal.
  The administration time is approximately 10 minutes. It is administered as a paper-and-pencil test, it can be conducted by healthcare professionals.
Change in physical, mental and social healths aspects related to quality of life | The first measurement time will be at the beginning of the study, the second at the end of the 10-week intervention, and the third a follow-up 4 weeks later.
  It will be measured with the Multiple Sclerosis Quality of Life-54 (MSQOL-54). It is a comprehensive health-related quality of life measure specifically designed for individuals with multiple sclerosis (MS). Evaluates the overall quality of life in MS patients, covering physical, mental, and social health aspects.
  Consists of 54 items, including 36 items from the SF-36 Health Survey and 18 additional items specific to MS. It generates 12 subscales and two summary scores.
  Subscales: Physical function, role limitations (physical and emotional), pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function.
  Summary Scores: Physical health composite and mental health composite. The administration time is approximately 11-18 minutes. It can be self-administered questionnaire, but can also be conducted as an interview if necessary.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Asociación Mostoleña de Esclerosis Múltiple (AMDEM), Móstoles, Madrid
  - Fundación Esclerosis Multiple Madrid (FEMM), Madrid

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of Individual Participant Data (IPD) has not yet been finalized. We are currently evaluating the potential benefits and risks associated with data sharing, including considerations related to patient privacy, data security, and the potential for future research collaborations. Our goal is to ensure that any decision made will maximize the scientific value of the data while protecting the rights and confidentiality of our participants. We will update our data sharing plans as soon as a decision is reached.